CLINICAL TRIAL: NCT01274962
Title: An Adaptative Randomized Phase II Study on the Timing of FOLFOX for Patients With Operable Stage III Rectal Cancer
Brief Title: A Study on the Timing of FOLFOX for Patients With Operable, Node Positive Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Dr. Te Vuong, Director Radiation Oncology Department, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KIR 009
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Operable T2-3N+M0 Rectal Cancer (Stage III)
MeSH Terms: interventions — Folfox protocol

ARMS (2):
- A - neoadjuvant chemotherapy (Experimental): Patients in arm A will receive 6 cycles of FOLFOX chemotherapy prior to radiotherapy and surgery as well as 6 cycles of chemotherapy in adjuvant
  Interventions: Drug: FOLFOX; Radiation: high dose rate endorectal brachytherapy
- Arm B - adjuvant chemotherapy (Experimental): Patients in arm B will receive 12 cycles of FOLFOX after radiotherapy and surgery
  Interventions: Drug: FOLFOX; Radiation: high dose rate endorectal brachytherapy

INTERVENTIONS:
Drug: FOLFOX — * Oxaliplatin* 85 mg/m2 IV in 500 mL of D5W over 120 minutes
  * Folinic Acid (Leucovorin)* 400 mg/m2 IV in 250 ml D5W over 120 minutes
  * 5-Fluorouracil (5-FU) 400 mg/m2 IV bolus, after Folinic Acid
  * 5-Fluorouracil** 2400 mg/m2 IV over 46 h in D5W to a total volume of 92 mL by continuous infusion at 2 mL/hour.
  * Repeat every 14 days for 6 cycles in the arm A and to be completed with 6 cycles after surgery and 12 cycles in arm B.
  If necessary the schedule may be modified +/- 3 days.
Radiation: high dose rate endorectal brachytherapy — High dose rate endorectal brachytherapy, consisting in a total dose of 26 Gy in 4 daily fractions of 6.5 Gy.

SUMMARY:
This study is proposed to evaluate whether giving part of the chemotherapy prior to radiotherapy and surgery (as opposed to standard of care, which involves giving all the chemotherapy after radiotherapy and surgery) for patients with node positive operable rectal cancer will result in higher patient compliance to chemotherapy.

DETAILED DESCRIPTION:
In recent randomized studies with preoperative combined chemotherapy and external beam radiation (EBRT/CT) with total mesorectal excision (TME surgery), the compliance to adjuvant chemotherapy ranged from 42.9% to 70%. This low compliance rate could influence the efficacy of chemotherapy. This is quite unique to patients with rectal cancer, since compliance is not a major issue in patients with colon cancer, belonging to the same age group. Therefore, it is reasonable to postulate that this difference might due to the additive toxicity burden of neoadjuvant EBRT/CT and TME.

In this randomized phase II study, compliance to chemotherapy will be compared in the two groups: In the first group, patients will receive half of their chemotherapy regimen in neoadjuvant and half in adjuvant; and, in the second group, patients will be receiving all their chemotherapy in adjuvant. Furthermore, brachytherapy will be used to deliver radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Pathology: Adenocarcinoma of the rectum.
2. T2 (CRM+) or T3 tumour at ≤ 10 cm from the A-V margin (as per MRI criteria)
3. Evidence of perirectal nodes on MRI or EUS (N1 or N2), any CRM+ and N0 tumor, or any EMVI+ tumor
4. Tumors with an adequate lumen to allow the positioning of the Oncosmart intracavitary mould applicator (e.g. non obstructive tumor).
5. Tumour of less than 3.5 cm thickness documented at the CT Simulator.
6. Patient should be a suitable candidate for surgery and chemotherapy.
7. WHO performance status 0-2
8. Age > 18 years.
9. Written informed consent.
10. Adequate birth control measures in women with childbearing potential.

Exclusion Criteria:

1. Patients with positive extramesorectal or pelvic nodes (e.g. iliac, lateral).
2. Evidence of distant metastases (M1).
3. Previous pelvic radiation.
4. Other cancers except for basal cell carcinoma of the skin or CIS of the cervix.
5. Presence of multiples small bowel loops trapped within the immediate tumor bed (post hysterectomy or prostatectomy).
6. Extension of malignant disease to the anal canal
7. Patients with severe co-morbid conditions (recent MI, infections, AIDS, etc)
8. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Compliance to chemotherapy - patients receiving at least 85% of planned full-dose of chemotherapy prescribed at each cycle for the 12 cycles | 1 year post diagnosis

SECONDARY OUTCOMES:
Disease free survival rate (local recurrence and metastases) | 5 years post surgery
Overall survival rate | 5 years post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Te Vuong, MD, Principal Investigator — Sir Mortimer B. Davis - Jewish General Hospital
Locations (8):
- Canada (8):
  - Hôpital de Gatineau, Gatineau, Quebec
  - Hôpital Charles LeMoyne, Greenfield Park, Quebec
  - Centre Hospitalier Pierre-Boucher, Longueuil, Quebec
  - CHUM-Hôpital St-Luc, Montreal, Quebec
  - Sir Mortimer B. Davis - Jewish General Hospital, Montreal, Quebec
  - Hôpital Honoré-Mercier, Saint-Hyacinthe, Quebec
  - Hôpital du Suroît, Salaberry-de-Valleyfield, Quebec
  - CHUQ - Hôtel-Dieu de Québec, Québec